CLINICAL TRIAL: NCT02827500
Title: Predischarge Initiation of Ivabradine in the Management of Heart Failure (PRIME-HF)
Acronym: PRIME-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071309
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Ivabradine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ivabradine (Active Comparator): Active Comparator: ivabradine
  Interventions: Drug: ivabradine
- usual care (Placebo Comparator): Placebo Comparator: usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Drug: ivabradine — Active Comparator: ivabradine
  Other Names: Corlanor
  Arms: ivabradine
Other: Usual Care — Placebo Comparator: usual care
  Arms: usual care

SUMMARY:
The PRIME-HF study is a multi-center, patient-level, randomized, open-label study of approximately 450 patients with reduced (left ventricular ejection fraction) LVEF of ≤ 35% and heart-rate ≥70 beats per minute (bpm) who are being discharged from the hospital following stabilization from acute heart failure (HF)(primary or secondary) and will be randomized to a treatment strategy of predischarge initiation of ivabradine or usual care.

All participants should have a follow-up visit within 7-14 days of hospital discharge. Heart rate and systolic blood pressure will be assessed at this clinical visit. For participants randomized to predischarge initiation of ivabradine and on ivabradine 5mg BID, the heart rate may be used to adjust the dose the dose to 2.5mg BID or 7.5mg BID. For participants randomized to usual care, ivabradine may be initiated at the provider's discretion. All participants will have a second follow-up study visit 6 weeks (42 +/- 14 days) post-discharge. Heart rate, systolic blood pressure and quality of life (KCCQ and PGA) will be assessed. For participants already taking ivabradine in either treatment group, the heart rate may again be used to adjust the dose of ivabradine. For participants not yet receiving ivabradine, it may be initiated at the provider's discretion. All participants will receive a 90 (+/-7) day post-discharge phone call by site to assess for event status and tolerability of ivabradine. All participants will have a final study visit at 180 (+/-14) days post-discharge. Heart rate, systolic blood pressure and quality of life (Kansas City Cardiomyopathy Questionnaire and Patient Global Assessment) will be assessed. The attending physician may initiate ivabradine per usual care clinical practice.

The primary hypothesis of the PRIME-HF study is that, compared with usual care, a treatment strategy of initiation of ivabradine prior to discharge for a hospitalization with acute HF will be associated with a greater proportion of participants using ivabradine at 180 days. Secondary objectives are to assess the impact of predischarge initiation of ivabradine on:Heart Rate (Change in heart rate from baseline to 180 days and Median heart rate at 180 days) and Patient-Centered Outcomes (Kansas City Cardiomyopathy Questionnaire (KCCQ) and Patient Global Assessment (PGA)). Tertiary objectives will be to explore the impact of predischarge initiation of ivabradine on other assessments of evidence-based implementation of ivabradine and beta-blockers at 180 days. Evaluations will incorporate data based on whether or not indication status was retained and whether or not an ivabradine prescription was provided. Tolerability of ivabradine and adverse events during study follow-up.

DETAILED DESCRIPTION:
* Purpose of the study The primary hypothesis of the PRIME-HF study is that, compared with usual care, a treatment strategy of initiation of ivabradine prior to discharge for a hospitalization with acute HF (primary or secondary) will be associated with a greater proportion of participants using ivabradine at 180 days. Secondary objectives are to assess the impact of predischarge initiation of ivabradine on:Heart Rate (Change in heart rate from baseline to 180 days and Median heart rate at 180 days) and Patient-Centered Outcomes (Kansas City Cardiomyopathy Questionnaire (KCCQ) and Patient Global Assessment (PGA)). Tertiary objectives will be to explore the impact of predischarge initiation of ivabradine on other assessments of evidence-based implementation of ivabradine and beta-blockers at 180 days. Evaluations will incorporate data based on whether or not indication status was retained and whether or not an ivabradine prescription was provided. Tolerability of ivabradine and adverse events during study follow-up will be assessed. Barriers to acquisition of ivabradine will be explored.
* Background & significance Heart failure is a major public health issue. More than 5 million Americans have HF and the prevalence is expected to increase as the population ages and survival from coronary, hypertensive, and valvular heart disease improves. Data from randomized clinical trials have established the efficacy of a number of medical and device therapies for patients with chronic Heart failure with reduced ejection fraction (HFrEF), but patient outcomes remain poor, especially after a hospitalization for heart failure. The 1-year mortality rate after a HF hospitalization is 20-30%, and this number has been relatively unchanged over the past decade. These data suggest that there is an unmet need for novel treatment strategies and supports the assessment of new approaches in the post-acute HF setting.

There is also wide variation in the implementation of clinical trial evidence into routine practice. Previous data highlight a multi-year gap between the generation of new evidence through clinical trials and the adoption of the data into routine clinical practice. This gap in care translates into many unnecessary deaths and hospitalizations each year for patients with HFrEF. While there are multiple reasons for this quality gap, clinical inertia has most often been noted as a major barrier. Ivabradine have been approved for use in Europe for several years for patients with symptomatic chronic HFrEF (LVEF <35%) and a heart rate >75 bpm on guideline-directed medical therapy (or intolerance/contra-indication to beta-blocker use). Ivabradine was recently approved for use in the United States. However, no US data exist regarding the potential adoption of ivabradine into routine clinical care.

Since ivabradine is a newly approved drug, this study also serves as a strategy trial to challenge study sites to explore drug acquisition for a drug that has been proven efficacious to the heart failure population and has been added to 2016 ACC/AHA/HFSA guidelines, however, has not been adopted rapidly into clinical practice. Ivabradine is not being provided for this study. Data are being captured to assess the number of subjects who were able to obtain ivabradine pre and post discharge as well as the barriers to acquisition.

Previous data for patients with HFrEF suggest that the hospital setting may provide a unique opportunity for patients to initiate guideline-directed medical therapy. In the Initiation Management Predischarge: Process for Assessment of Carvedilol Therapy in HF (IMPACT-HF) study, patients with an LVEF<40% hospitalized for HF that were started on carvedilol prior to hospital discharge were more likely to be on a beta-blocker at 60 days post-randomization compared to those receiving usual care. These improvements in care were achieved without increasing side effects or index hospitalization length of stay. Similar to beta-blockers and other medical therapies for HF, ivabradine was initially studied in patients with chronic HF. The initiation of ivabradine specifically in patients following stabilization for acute HF has not been evaluated.

• Design & procedures The PRIME-HF study is a multi-center, patient-level, randomized, open-label study of approximately 450 patients with reduced LVEF of ≤35% and heart-rate ≥70 bpm who are being discharged from the hospital following stabilization from acute HF and will be randomized to a treatment strategy of predischarge initiation of ivabradine or usual care.

All participants should have a follow-up visit within 7-14 days of hospital discharge. Heart rate and systolic blood pressure will be assessed at this clinical visit. For participants randomized to predischarge initiation of ivabradine and on ivabradine 5mg BID, the heart rate may be used to adjust the dose the dose to 2.5mg BID or 7.5mg BID. For participants randomized to usual care, ivabradine may be initiated at the provider's discretion. All participants will have a second follow-up study visit 6 weeks (42 +/- 14 days) post-discharge. Heart rate, systolic blood pressure and quality of life (KCCQ and PGA) will be assessed. For participants already taking ivabradine in either treatment group, the heart rate may again be used to adjust the dose of ivabradine. For participants not yet receiving ivabradine, it may be initiated at the provider's discretion. All participants will receive a 90 (+/-7) day post-discharge phone call by site to assess for event status and tolerability of ivabradine. All participants will have a final study visit at 180 (+/-14) days post-discharge. Heart rate, systolic blood pressure and quality of life (KCCQ and PGA) will be assessed. The attending physician may initiate ivabradine per usual care clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with acute HF (primary or secondary diagnosis) based on clinician assessment
2. A prior clinical diagnosis of HF (i.e., not a new diagnosis of heart failure during the current hospitalization)
3. Most recent LVEF ≤ 35% and within 6 months of randomization or LVEF ≤ 25% within 12 months of randomization
4. On optimal guideline-directed medical therapy for HFrEF (or previously deemed intolerant) as determined by the clinician including ACE-inhibitors or angiotensin receptor antagonists or neprilysin inhibition, aldosterone receptor antagonists, and maximally-tolerated doses of beta-blockers at the time of current evaluation (which may differ from long-term targets)

   * Maximally-tolerated doses of beta-blockers will be defined by the treating physician when considering aspects such as current dose relative to the target dose used in clinical trials, patient heart rate and blood pressure, and patient symptoms
   * Patients with intolerance or contraindication to beta-blocker use are eligible for enrollment (details will be documented in the case report form)
5. Age >18 years
6. Willingness to provide informed consent from the subject (or their guardian or legally authorized representative [LAR])
7. On the day of planned randomization, all participants:

   * Must be in sinus rhythm with a resting heart rate >70 bpm as measured on ECG or 10-second rhythm strip
   * Must have a blood pressure of >90/50 mm Hg

Exclusion Criteria:

1. Documented plan for uptitration of beta-blocker in the following 4 weeks
2. Permanent atrial fibrillation or atrial flutter
3. Patients with recent atrial fibrillation or flutter defined by either precipitating the current HF hospitalization or occurring during the current HF hospitalization
4. History of untreated sick sinus syndrome, sinoatrial block, or second and third degree atrio-ventricular block
5. Pacemaker with atrial or ventricular pacing (except biventricular pacing) >40% of the time
6. Family history or congenital long QT syndrome
7. Recent myocardial infarction (<2 months prior to screening) [troponin elevation secondary to acute HF as determined by the clinician is not an exclusion]
8. Acute or chronic severe liver disease as evidenced by any of the following: encephalopathy, variceal bleeding, INR > 1.7 in the absence of anticoagulation treatment
9. Creatinine clearance <15 mL/min within 48 hours of screening that was not due to acute kidney injury that resolved
10. Planned mechanical circulatory support within 180 days
11. Pregnant or breastfeeding women. Women with child-bearing potential should use effective contraception.
12. Medical conditions likely to lead to poor non-cardiac survival at 180 days (e.g., cancer)
13. Inability to comply with planned study procedures
14. If the following medications are needed at inclusion or during the study:

    * Non-dihydropyridine calcium channel blockers (e.g., diltiazem and verapamil)
    * Class I anti-arrhythmics (e.g., quinidine, procainamide, lidocaine, phenytoin)
    * Strong inhibitors of cytochrome P450 3A4 (CYP3A4), including some macrolide antibiotics (e.g., clarithromycin, erythromycin), cyclosporine, antiretroviral drugs (e.g., ritonavir, nelfinavir), and systemic azole antifungal agents (e.g., ketoconazole, itraconazole), and nefazodone
    * Inducers of cytochrome P450 3A4 (CYP3A4) including St. John's wort, rifampicin, barbiturates, and phenytoin.
    * Treatments known to be associated with significant prolongation of the QT interval, including sotalol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2016-07; Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Mentz, MD, Principal Investigator — Duke Clinical Research Institute
Locations (20):
- United States (20):
  - University of Colorado at Denver and Health Sciences Center, Aurora, Colorado
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Athens Regional Medical Center, Athens, Georgia
  - University Hospital, Augusta, Georgia
  - Tanner Medical Center, Carrollton, Georgia
  - Midwest Cardiovascular Research, Elkhart, Indiana
  - Saint Vincent Medical Group, Inc., Indianapolis, Indiana
  - Great Lakes Heart Center of Alpena, Alpena, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New York Methodist Hospital, Brooklyn, New York
  - Mount Sinai Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University- Davis Heart and Lung Research Institute, Columbus, Ohio
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - William Beaumont Army Medical Center, El Paso, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin

REFERENCES:
- [Derived] Mentz RJ, DeVore AD, Tasissa G, Heitner JF, Pina IL, Lala A, Cole RT, Lanfear DD, Patel CB, Ginwalla M, Old W, Salacata AS, Bigelow R, Fonarow GC, Hernandez AF. PredischaRge initiation of Ivabradine in the ManagEment of Heart Failure: Results of the PRIME-HF Trial. Am Heart J. 2020 May;223:98-105. doi: 10.1016/j.ahj.2019.12.024. Epub 2020 Feb 28. PMID 32217365

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects hospitalized with acute heart failure were randomized prior to discharge from September 2016- April 2018.
Groups:
- Pre-discharge Ivabradine: Active Comparator: ivabradine
  ivabradine: Active Comparator: ivabradine
Period: Overall Study
Arm/Group | Usual Care | Pre-discharge Ivabradine
Started | 52 | 52
Completed | 33 | 45
Not Completed | 19 | 7
Not completed — Death | 7 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Missing primary endpoint data | 3 | 1
Not completed — Other | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Pre-discharge Ivabradine | Total
Number analyzed (Participants) | 52 | 52 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (12) | 56.5 (14.8) | 57.5 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 14 | 37
  Male | 29 | 38 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 12
  Not Hispanic or Latino | 46 | 41 | 87
  Unknown or Not Reported | 0 | 5 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 34 | 33 | 67
  White | 17 | 17 | 34
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 52 | 52 | 104

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Taking Ivabradine at 180 Days
Time Frame: 180 days
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 52 | 52
Participants | 6 | 21
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; Test type: Superiority; p = 0.002, Regression, Logistic; Odds Ratio, log = 5.19, 95% CI 2-sided [1.88 to 14.33]

2. Secondary Outcome: Change in Heart Rate
Description: Change from baseline is calculated as 180 days - baseline results. Heart rate results are obtained from vital sign assessment when available otherwise results from ECG assessment are used.
Time Frame: baseline,180 days
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 52 | 52
beats per minute | -10.2 (20.6) | 0.9 (16.7)
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; Test type: Superiority; p = 0.011, Regression, Linear

3. Secondary Outcome: Heart Rate at 180 Days
Description: Heart rate results are obtained from vital sign assessment when available otherwise results from ECG assessment are used from day 180.
Time Frame: 180 days
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 52 | 52
beats per minute | 85.4 (16.7) | 77.2 (16.9)
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; The null hypothesis tested was that there is no difference in change in heart rate between the treatment arms; Test type: Superiority; p = 0.011, Regression, Linear

4. Secondary Outcome: Number of Patients With Heart Rate <70 Bpm at 180 Days
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 52 | 52
Participants | 11 | 20
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; The null hypothesis tested was that there is no difference between the treatment arms in the proportion of patients with heart rate < 70 BPM; Test type: Superiority; p = 0.054, Chi-squared, Corrected — The apriori threshold for statistical significance is alpha=0.05; The p-value is obtained using the F-test (combination of Chi-Squared tests) due to multiple imputation

5. Secondary Outcome: Changes in Symptoms and Quality of Life as Measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) Overall Summary Score
Description: Change from baseline is calculated as 180 day - baseline results. Scores range 0-100, where a higher score indicates a better outcome.
Time Frame: baseline, 180 days
Population: Participants who completed the KCCQ at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 29 | 38
score on a scale | 25.1 (23.9) | 23.2 (32)
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; Test type: Superiority; p = 0.717, Regression, Linear

6. Secondary Outcome: Changes in Symptoms and Quality of Life as Measured by Patient Global Assessment (PGA)
Description: Change from baseline is calculated as 180 day - baseline results. Scores range 0-100, where a higher score indicates a worse outcome.
Time Frame: baseline, 180 days
Population: Participants who completed the PGA at both timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Usual Care | Pre-discharge Ivabradine
Number analyzed (Participants) | 29 | 38
score on a scale | 13 (26) | 14.8 (29.4)
Statistical Analysis 1: Comparison: Usual Care vs Pre-discharge Ivabradine; Test type: Superiority; p = 0.784, Regression, Linear

ADVERSE EVENTS:
Time Frame: Events through day 194 (6 month +/- 2 week window)
Description: Only events of interest, serious and unexpected events, and events related to ivabradine use in the opinion of the site investigators were collected.
Arm/Group | Usual Care | Pre-discharge Ivabradine
All-Cause Mortality (participants affected / at risk) | 7/52 | 3/52
Serious Adverse Events (participants affected / at risk) | 2/52 | 3/52
Other Adverse Events (participants affected / at risk) | 10/52 | 1/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=52) | Pre-discharge Ivabradine (N=52)
Toxic Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular Fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=52) | Pre-discharge Ivabradine (N=52)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperhydrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT02827500/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02827500/SAP_001.pdf